CLINICAL TRIAL: NCT01205685
Title: A Phase II Trial of Endocrine Therapy in Combination With OSI-906 (an IGF-1R Inhibitor) and Erlotinib (Tarceva®, an EGFR Inhibitor) in Patients With Hormone-sensitive Metastatic Breast Cancer
Brief Title: Endocrine Therapy + OSI-906 With or Without Erlotinib for Hormone-Sensitive Metastatic Breast Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: PI closed study early, all patients experienced severe toxicities and progressed
Sponsor: Vanderbilt-Ingram Cancer Center (Other)
Responsible Party: Principal Investigator, Ingrid Mayer, MD, Assistant Professor of Medicine; Clinical Director, Breast Cancer Program; Medical Oncologist, Vanderbilt-Ingram Cancer Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: VICC BRE 09112
Record Dates: First submitted 2010-09-17; First posted 2010-09-20 (Estimated); Results first posted 2012-09-11 (Estimated); Last update posted 2012-09-11 (Estimated); Status verified 2012-08

CONDITIONS: Hormone-sensitive Metastatic Breast Cancer
MeSH Terms: interventions — 3-(8-amino-1-(2-phenylquinolin-7-yl)imidazo(1,5-a)pyrazin-3-yl)-1-methylcyclobutanol; Erlotinib Hydrochloride; Letrozole; Goserelin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- OSI-906 + Erlotinib + Letrozole + Goserelin (Experimental): * OSI-906 in a pill form, by mouth, twice a day (12 hours a part)
  * Erlotinib in a pill form, by mouth, once a day
  * Letrozole in a pill form, by mouth, once a day
  * Goserelin, by injection once per month for women who are pre-menopausal
  Interventions: Drug: OSI-906; Drug: Erlotinib; Drug: Letrozole; Drug: Goserelin

INTERVENTIONS:
Drug: OSI-906 — In a pill form by mouth, twice a day (12 hours apart)
  During the safety run portion of the study"
  * Dose level 2 = 150 mg twice a day
  * Dose level 1 = 100 mg twice a day
  * Dose level -1 = 100 mg twice a day
  * Dose level -2 = 100 mg twice a day
Drug: Erlotinib — During the safety run phase of the study:
  * Dose Level 2 = 100 mg/d
  * Dose Level 1 = 100 mg/d
  * Dose Level -1= 75 mg/d
  * Dose Level -2 = 50 mg/d
Drug: Letrozole — In a pill form, by mouth, once per day at 2.5 mg/d.
Drug: Goserelin — For pre-menopausal patients only. Given as an injection once a month at 3.6 mg/month.

SUMMARY:
Erlotinib attacks a part of cancer cells that helps them live and grow. Studies done in human beings show that this drug can make a difference in the way anti-estrogens work in hormone-sensitive breast cancers. OSI-906 attacks a different part of the cancer cell that helps them live and grow. Studies done in the laboratory show that OSI-906 can make a difference in the way anti-estrogens work in hormone-sensitive breast cancers.

DETAILED DESCRIPTION:
The safety run component of this trial is to determine the safety profile of the OSI-906, erlotinib and anti-endocrine treatment combination. The phase II component evaluates the antitumor activity of the combination OSI-906, erlotinib and endocrine therapy.

ELIGIBILITY:
Inclusion Criteria:

* Patients must provide informed written consent.
* Patients must be ≥18 years of age.
* ECOG performance status 0-1.
* Patients with clinical stage IV invasive mammary carcinoma, previously documented by histological analysis, which is ER-positive and/or PR-positive by immunohistochemistry (IHC), which had previous endocrine therapy in the metastatic setting or had metastatic recurrence within 6 months of adjuvant endocrine therapy. Patients may have either measurable or non-measurable disease, both are allowed.
* Patients whose breast cancers are also HER2-overexpressed (IHC 3+ or FISHpositive) need to have had previous treatment exposure to trastuzumab (Herceptin®)
* Life expectancy ≥ 6 months
* Patients must have adequate hematologic, hepatic, and renal function. All tests must be obtained less than 2 weeks from study entry. This includes:

  * ANC ≥1250/mm3
  * Platelet count ≥100,000/mm3
  * Creatinine ≤1.5X upper limits of normal
  * Bilirubin, SGOT, SGPT ≤ 1.5 X upper limits of normal if no liver metastasis present*
  * Bilirubin, SGOT, SGPT, alkaline phosphatase ≤ 3 X upper limits of normal if liver metastasis present* *for patients with Gilbert's syndrome, direct bilirubin will be measured instead of total bilirubin
* Able to swallow and retain oral medication.
* Pre-menopausal patients must have a negative pregnancy test prior to participating in the study. Women of childbearing age and their male counter parts should use a barrier method of contraception during and for 3 months following protocol therapy.
* Post-menopausal female subjects should be defined prior to protocol enrollment by any of the following:

  * Subjects at least 55 years of age;
  * Subjects under 55 years of age and amenorrheic for at least 12 months or follicle-stimulating hormone (FSH) values ≥40 IU/L and estradiol levels

    ≤20 IU/L;
  * Prior bilateral oophorectomy or prior radiation castration with amenorrhea for at least 6 months.
* Patients may receive concurrent radiation therapy to painful bone metastases or areas of impending bone fracture as long as radiation therapy is initiated prior to study entry. Patients who have received prior radiotherapy must have recovered from any toxicity induced by this treatment (toxicity grade ≤ 1).
* Patients must be disease-free of prior invasive cancers for > 5 years with the exception of basal or squamous cancer of the skin or cervical carcinoma in situ.
* Subjects must complete all screening assessments as outlined in the protocol.
* Patients must have available tissue (archived formalin-fixed paraffin embedded blocks (FFPB) or fresh frozen tissue from original diagnosis or metastatic setting)for correlative studies. Tissue needs to be sent to VUMC (see Appendix E) at the time of registration. Patients will not be able to start study drugs without tissue availability.

Exclusion Criteria:

* Locally recurrent resectable breast cancer.
* Pregnant or lactating women.
* Patients must not have had > than 4 prior chemotherapy treatments in the metastatic setting. This restriction does not include endocrine therapies or single agent biologic therapies.
* Use of CYP3A4 and CYP1A2 modifiers or drugs that prolong QTcF with high risk for Torsade de Pointes (see Appendix A)
* Any kind of malabsorption syndrome significantly affecting gastrointestinal function.
* History of other malignancy within 5 years prior to enrollment. Subjects with a history of completely resected non-melanoma skin cancer or successfully treated in situ carcinomas are eligible.
* Patients with baseline QTcF> 450 msec
* Patients with diabetes, glucose > 160 mg/dL or receiving ongoing antihyperglycemic therapies
* Uncontrolled intercurrent illness including, but not limited to:

  * ongoing or active infection requiring parenteral antibiotics
  * impairment of lung function (COPD > grade 2, lung conditions requiring oxygen therapy)
  * symptomatic congestive heart failure (class III or IV of the New York Heart Association classification for heart disease)
  * unstable angina pectoris, angioplasty, stenting, or myocardial infarction within 6 months
  * uncontrolled hypertension (systolic blood pressure >180 mm Hg or diastolic blood pressure >100 mm Hg, found on two consecutive measurements separated by a 1-week period despite adequate medical support)
  * clinically significant cardiac arrhythmia (multifocal premature ventricular contractions, bigeminy, trigeminy, ventricular tachycardia that is symptomatic or requires treatment [National Cancer Institute -Common Terminology Criteria for Adverse Events, Version 4.0, grade 3]
  * psychiatric illness/social situations that would compromise patient safety or limit compliance with study requirements including maintenance of a compliance/pill diary
* Patients with symptomatic brain metastases (patients with a history of brain metastases must be clinically stable for more than 3 weeks from completion of radiation treatment and not taking steroids or therapeutic anticonvulsants that are CYP3A4 modifiers)
* Patients with asymptomatic brain metastasis on prophylactic anticonvulsants that are CYP3A4 modifiers
* Concurrent anti-cancer therapy (chemotherapy, radiation therapy, surgery, immunotherapy, hormonal therapy, biologic therapy) other than the ones specified in the protocol. Patients must have discontinued the above cancer therapies for 1 week prior to the first dose of study medication, as well as recovered from toxicity (to ≤ than grade 1, except for alopecia, neuropathy, and ANC, which should be ≥ 1250/mm3) induced by previous treatments. Any other investigational drugs should be discontinued 2 weeks prior to the first dose of study medication.
* Prior therapy with an IGF-1R inhibitor

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2010-05; Primary Completion 2011-07 (Actual); Study Completion 2011-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ingrid Mayer, M.D., Principal Investigator — Vanderbilt-Ingram Cancer Center
Locations (3):
- United States (3):
  - Vanderbilt-Ingram Oncology Cool Springs, Franklin, Tennessee
  - Vanderbilt One Hundre Oaks, Nashville, Tennessee
  - Vanderbilt-Ingram Cancer Center, Nashville, Tennessee

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted from May 2010 and closed early one year later, May 2011.
Pre-assignment Details: 12 patients consented, one of which was determined to be ineligible.
Period: Overall Study
Arm/Group | OSI-906 + Erlotinib + Letrozole + Goserelin
Started | 11
Completed | 0
Not Completed | 11
Not completed — Disease Progression | 10
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Arm/Group | OSI-906 + Erlotinib + Letrozole + Goserelin
Number analyzed (Participants) | 11
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 8
  >=65 years | 3
Age Continuous [Mean (Standard Deviation); unit: years] | 59 (1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11
  Male | 0
Region of Enrollment [Number; unit: participants]
  United States | 11

OUTCOME MEASURES:

1. Primary Outcome: Anti-tumor Activity of OSI-906
Description: Time to progression measured in months from study entry to date of disease progression
Time Frame: From study entry to 6 months
Population: Patients who received treatment and who were available for determination of disease progression. One patient withdrew after beginning of treatment and was not available for determination of the duration of disease progression.
Measure: Median (Full Range); unit: months
Arm/Group | OSI-906 + Erlotinib + Letrozole + Goserelin
Number analyzed (Participants) | 10
months | 2 [0 to 2]

2. Secondary Outcome: Safety Profile Based on Number of Patients With Each Worst-grade Toxicity
Description: According to National Cancer Institute Common Toxicity Criteria for Adverse Events with 1 = mild, 2 = moderate, 3 = severe, 4 = life threatening/disabling, and 5 = death.
Time Frame: Every 4 weeks up to 24 weeks
Population: Patients who received treatment and experienced an adverse event.
Measure: Number; unit: participants
Arm/Group | OSI-906 + Erlotinib + Letrozole + Goserelin
Number analyzed (Participants) | 11
participants
  Patients with worst grade toxicity of 1 | 2
  Patients with worst grade toxicity of 2 | 6
  Patients with worst grade toxicity of 3 | 3
  Patients with worst grade toxicity of 4 | 0
  Patients with worst grade toxicity of 5 | 0

3. Secondary Outcome: Number of Participants With Tumor Response Per RECIST
Description: Per RECIST criteria v. 1.1: measurable lesions: complete response (CR) disappearance of target lesions, partial response (PR) > 30% decrease in the sum of the longest diameter (LD) of target lesions, progressive disease (PD) > 20% increase in the sum of the LD of target lesions or appearance of new lesions, stable disease (SD) neither sufficient decrease nor increase of the sum of smallest sum of the LD of target lesions
Time Frame: Every 12 weeks to tumor progression
Population: Patients who were available for measurement of tumor response.
Measure: Number; unit: participants
Arm/Group | OSI-906 + Erlotinib + Letrozole + Goserelin
Number analyzed (Participants) | 10
participants
  Complete Response | 0
  Partial Response | 0
  Stable Disease | 0
  Progressive disease | 10

4. Secondary Outcome: Correlative Studies
Description: Biomarkers associated with response to OSI-906 + Erlotinib + Letrozole + Goserelin
Time Frame: < or = to 2 weeks before initiation of Phase II study treatment period
Population: No correlative studies were performed because the study did not move to the Phase II portion
Arm/Group | OSI-906 + Erlotinib + Letrozole + Goserelin
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Arm/Group | OSI-906 + Erlotinib + Letrozole + Goserelin
Serious Adverse Events (participants affected / at risk) | 2/11
Other Adverse Events (participants affected / at risk) | 11/11
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | OSI-906 + Erlotinib + Letrozole + Goserelin (N=11)
Acute kidney injury (Renal and urinary disorders) | 1 (1)
Hypercalcemia (Metabolism and nutrition disorders) | 2 (2)
Fatigue (General disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | OSI-906 + Erlotinib + Letrozole + Goserelin (N=11)
alanine aminotransferase increased (Investigations) | 4 (7)
alkaline phosphatase increased (Investigations) | 3 (4)
anemia (Blood and lymphatic system disorders) | 3 (5)
anorexia (Metabolism and nutrition disorders) | 1 (1)
aspartate aminotransferase increased (Investigations) | 5 (5)
back pain (Musculoskeletal and connective tissue disorders) | 1 (1)
bladder spasm (Renal and urinary disorders) | 1 (1)
creatinine increased (Investigations) | 1 (3)
depression (Psychiatric disorders) | 2 (2)
diarrhea (Gastrointestinal disorders) | 4 (4)
dizziness (Nervous system disorders) | 1 (1)
dry eye (Eye disorders) | 1 (1)
dry mouth (Gastrointestinal disorders) | 1 (1)
dry skin (Skin and subcutaneous tissue disorders) | 2 (2)
electrocardiagram QT interval prolonged (Cardiac disorders) | 2 (2)
epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (2)
eye disorders (Eye disorders) | 1 (2)
hypercalcemia (Metabolism and nutrition disorders) | 2 (5)
hyperglycemia (Metabolism and nutrition disorders) | 5 (5)
hypocalcemia (Metabolism and nutrition disorders) | 2 (2)
hypoglycemia (Metabolism and nutrition disorders) | 1 (1)
hypokalemia (Metabolism and nutrition disorders) | 4 (5)
hyponatremia (Metabolism and nutrition disorders) | 3 (4)
insomnia (Psychiatric disorders) | 1 (1)
leukocytosis (Blood and lymphatic system disorders) | 1 (11)
mucositis oral (Gastrointestinal disorders) | 2 (2)
nausea (Gastrointestinal disorders) | 2 (2)
non-cardiac chest pain (Musculoskeletal and connective tissue disorders) | 1 (1)
pain (General disorders) | 1 (1)
rash acneiform (Skin and subcutaneous tissue disorders) | 7 (8)
rash macro-papular (Skin and subcutaneous tissue disorders) | 1 (1)
skin and subcutaneous tissue disorders Other (Skin and subcutaneous tissue disorders) | 1 (1)
upper respiratory infection (Respiratory, thoracic and mediastinal disorders) | 1 (1)
urinary incontinence (Renal and urinary disorders) | 1 (1)
flu-like symptoms (General disorders) | 1 (1)
fatigue (General disorders) | 2 (3)
pruritis (Skin and subcutaneous tissue disorders) | 1 (1)
gastrointestinal disorders Other (Gastrointestinal disorders) | 1 (1)
general disorders and administrative site disorders-other (General disorders) | 1 (2)
hypothyroidism (Endocrine disorders) | 1 (1)
pain-bone (Musculoskeletal and connective tissue disorders) | 1 (1)
flu-like symptoms (General disorders) | 1 (1)
neutrophil count decreased (Investigations) | 1 (1)
white blood cells decreased (Investigations) | 1 (1)
leukocytosis (Blood and lymphatic system disorders) | 1 (1)
acute kidney injury (Renal and urinary disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes